CLINICAL TRIAL: NCT01159860
Title: Is Cryosurgery or Curettage More Effective at Treating Seborrheic Keratoses?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Milton S. Hershey Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: IRB Protocol No. 33895
Record Dates: First submitted 2010-07-09; First posted 2010-07-12 (Estimated); Last update posted 2018-05-25 (Actual); Status verified 2018-05

CONDITIONS: Seborrheic Keratosis
Keywords: seborrheic keratoses; cryosurgery; curettage
MeSH Terms: conditions — Keratosis, Seborrheic | interventions — Cryosurgery; Curettage

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cryosurgery (Active Comparator): One lesion on the patients' trunk or proximal extremities will be treated with cryosurgery.
  Interventions: Procedure: cryosurgery
- Curettage (Active Comparator): One lesion on one side of the patients' trunk or proximal extremities will be treated by curettage.
  Interventions: Procedure: Curettage

INTERVENTIONS:
Procedure: cryosurgery — freezing of lesion with liquid nitrogen
  Arms: Cryosurgery
Procedure: Curettage — the lesion will be anesthetized and destroyed with a curette.
  Arms: Curettage

SUMMARY:
Seborrheic keratoses (SK's) are very common, but harmless skin lesions that commonly appear during adult life. Patients with seborrheic keratoses frequently desire treatment due to symptoms of itching and irritation or for cosmetic purposes. Seborrheic keratoses can be easily removed and have been treated in a number of different ways. Two of the simplest and most successful ways to remove seborrheic keratoses are cryosurgery and curettage.

The investigators are conducting this study to see which of these two treatments has the best result.

Approximately 24-30 people will take part in this research study at the Hershey Medical Center.

ELIGIBILITY:
Inclusion Criteria:

* have at least 1 seborrheic keratosis on each side of his/her trunk or proximal extremities.
* be able to understand the consent form and evaluation of treatment questionnaire.

Exclusion Criteria:

* Children <18 are excluded from this study based on their inability to independently complete the informed consent and research associated questionnaire.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2010-07; Primary Completion 2012-05-11 (Actual); Study Completion 2013-06-06 (Actual)

PRIMARY OUTCOMES:
Partial or complete resolution of treated lesion. | 6 weeks
  Follow up evaluation by a blinded physician along with the gathering of patient information via questionnaires will be obtained at the completion of the study.

CONTACTS AND LOCATIONS:
Overall Officials: Lance D. Wood, M.D., Principal Investigator — Milton S. Hershey Medical Center
Locations (1):
- Penn State Milton S. Hershey Medical Center, Hershey, Pennsylvania, United States

REFERENCES:
- [Background] Brodsky J. Management of benign skin lesions commonly affecting the face: actinic keratosis, seborrheic keratosis, and rosacea. Curr Opin Otolaryngol Head Neck Surg. 2009 Aug;17(4):315-20. doi: 10.1097/MOO.0b013e32832d75e3. PMID 19465852
- [Background] Herron MD, Bowen AR, Krueger GG. Seborrheic keratoses: a study comparing the standard cryosurgery with topical calcipotriene, topical tazarotene, and topical imiquimod. Int J Dermatol. 2004 Apr;43(4):300-2. doi: 10.1111/j.1365-4632.2004.02282.x. PMID 15090020